CLINICAL TRIAL: NCT06768879
Title: Sonographic Evaluation Of Uterine Fibroids At Different Locations In Patient With Irregular Menstrul Cycle
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/033
Record Dates: First submitted 2024-12-18; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Menstrual Irregularity
MeSH Terms: conditions — Menstruation Disturbances | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Ultrasound — To evaluate the different location of uterine fibroids in patient with disturbed menstrual cycle on ultrasound

SUMMARY:
Uterine fibroids are a major cause of illness in women of a reproductive age. There are many factors involved in the growth and reduction of these common tumors. The most likely cause of fibroids is their effect on a woman's menstrual cycle. For accurate diagnosis numerous diagnostic markers on ultrasound are present which increases the efficacy of ultrasound to diagnose uterine fibroids.

DETAILED DESCRIPTION:
To evaluate the different location of uterine fibroids in patient with disturbed menstrual cycle on Ultrasound.

The descriptive and cross-sectional study was conducted. A total of 97 patient data were collected. All the patients with uterine fibroids due to heavy bleeding, abdominal pain, pelvic pain, disturbance in menstrual cycle undergoing ultrasound were included.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Pelvic pain
* Patient with Abdominal pain
* Patient with heavy bleeding
* Patient with Dysmenorrhea
* Polymenorrhea

Exclusion Criteria:

* Patient with H/O Cystectomy
* Patient with H/O cyst

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Irregular Menstrul Cycle
Study Population: Aim is to check Irregular Menstrul Cycle with Sonographic Evaluation Of Uterine Fibroids
Sampling Method: Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
two-dimensional ultrasound scan (GE Loginq P7 convex probe.3.5-5MHz) | 12 Months
  On ultrasound using (GE Loginq P7 convex probe.3.5-5MHz), a uterine fibroid is classically characterized as a solid, round, well-defined, hypoechoic, heterogeneous lesion within the myometrium, often showing acoustic shadowing at the edge of the lesion

CONTACTS AND LOCATIONS:
Locations (1):
- THQ hospital Pattoki/ Siddique medical center Pattoki, Pattoki, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No